CLINICAL TRIAL: NCT06479798
Title: Accuracy of Convex Probe EBUS-TBNA Versus FDG-PET/CT Imaging in Diagnosis of Suspected Lung Cancer & Staging of Concurrent Mediastinal Lymphadenopathy at Ain-Shams University Hospitals
Brief Title: Accuracy of Convex Probe EBUS-TBNA Versus FDG-PET/CT Imaging in Diagnosis and Staging of Lung Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Fatma Alzahraa, Assistant lecturer of pulmonology, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: department of chest diseases
Record Dates: First submitted 2024-06-22; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Lung Malignancies; Mediastinal Lymphadenopathy
Keywords: FDG-PET/CT; lung cancer; lung staging; EBUS-TBNA; mediastinal lymphadenopathy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This prospective, interventional cohort research was performed on 40 cases with suspected lung malignancies. All cases were examined via FDG-PET/CT followed by convex probe EBUS-TBNA for diagnosis of suspected lung cancer & staging of concurrent mediastinal lymphadenopathy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FDG PET and EBUS TBNA arm (Other): It is a single arm in which all patients undergo FDG PET and EBUS-TBNA
  Interventions: Diagnostic Test: Endo bronchial ultrasound transbronchial needle aspiration(EBUS-TBNA)

INTERVENTIONS:
Diagnostic Test: Endo bronchial ultrasound transbronchial needle aspiration(EBUS-TBNA) — Endo bronchial ultrasound enables visualization of parabronchial structures throughout a bronchoscopic procedure. EBUS-TBNA, which is considered a less invasive diagnostic tool for nodal staging compared to mediastinoscopy, allows real-time, direct sampling of hilar & MLNs under sonograghic guidance with concurrent cytological and histopathological examination
  Other Names: FDG-PET/CT

SUMMARY:
Lung cancer is a prevalent cause of cancer-related mortality on a global scale. Appropriate staging of lung cancer is of paramount importance, as it customizes treatment and predicts prognosis. Fludeoxyglucose-18 (FDG) positron emission tomography (PET) combined with low dose contrast computed tomography (CT) and endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) are two diagnostic modalities widely used in the field of staging & diagnosis of lung malignancies, the former depends on image analysis while the later enables real-time sampling of lymph nodes under sonographic guidance with concurrent cytological examination. The present research aims to compare the diagnostic and staging accuracies of (EBUS-TBNA) versus FDG-PET /CT as two diagnostic modalities in patients with suspected lung malignancies. However as a secondary outcome this study aims at monitoring the possible complications arising post EBUS-TBNA procedure.

DETAILED DESCRIPTION:
Lung cancer is a prevalent cause of cancer-related mortality on a global scale. Appropriate staging of lung cancer is of paramount importance, as it customizes treatment and predicts prognosis. Fludeoxyglucose-18 (FDG) positron emission tomography (PET) combined with low dose contrast computed tomography (CT) and endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) are two diagnostic modalities widely used in the field of staging & diagnosis of lung malignancies, the former depends on image analysis while the later enables real-time sampling of lymph nodes under sonographic guidance with concurrent cytological examination.

Objective: To compare the diagnostic and staging accuracy of convex probe EBUS-TBNA versus FDG - PET/CT as two diagnostic modalities in diagnosis of suspected lung cancer & staging of concurrent mediastinal lymphadenopathy Patients and Methods: This prospective, interventional cohort research was performed on 40 cases with suspected lung malignancies. All cases were examined via FDG-PET/CT followed by convex probe EBUS-TBNA for diagnosis of suspected lung cancer & staging of concurrent mediastinal lymphadenopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or more.
* Patients presented with centrally located suspiciously malignant lung masses with or without lymphadenopathy.
* patients with mediastinal lymphadenopathy only as evident by contrast - enhanced CT scan of the chest.
* patients with peripheral lung malignancy and mediastinal lymphadenopathy who were referred for MLN staging were also recruited to the research

Exclusion Criteria:

* All patients who were who were unfit for bronchoscopy as per international guidelines for practice.
* Cases are diagnosed with stage IV (metastatic) lung cancer.
* Patients with histopathological diagnosis other than malignancy (as Sarcoidosis, Tuberculosis).
* patients unfit for FDG-PET G-PET/CT examination (uncontrolled Hyperglycemia, renal impairment).
* Patients who refused to participate to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Comparing the diagnostic accuracies of both EBUS TBNA and FDG-PET /CT | 2 years
  Comparing the diagnostic yield of both modalies as they are considered primary main diagnostic and staging modalities for lung malignancies
Comparing the staging accuracies of both convex probe EBUS-TBNA versus FDG - PET/CT | 2 years
  Accurate staging of lung malignancies is considered crucial in determining the prognosis and specifying the treatment plan.

SECONDARY OUTCOMES:
Determine the complications | 2 years
  EBUS TBNA is a minimally invasive procedure having a very low rate of complications compared to mediastinoscopy, this study aims to monitor complications (if present)

CONTACTS AND LOCATIONS:
Overall Officials: Emad Korraa, MD, Study Director — Department of chest diseases and head of the bronchoscopy unit
Locations (1):
- Department of chest diseases , faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sehgal IS, Agarwal R, Dhooria S, Prasad KT, Aggarwal AN. Role of EBUS TBNA in Staging of Lung Cancer: A Clinician's Perspective. J Cytol. 2019 Jan-Mar;36(1):61-64. doi: 10.4103/JOC.JOC_172_18. PMID 30745743
- [Background] Kuo CH, Chen HC, Chung FT, Lo YL, Lee KY, Wang CW, Kuo WH, Yen TC, Kuo HP. Diagnostic value of EBUS-TBNA for lung cancer with non-enlarged lymph nodes: a study in a tuberculosis-endemic country. PLoS One. 2011 Feb 25;6(2):e16877. doi: 10.1371/journal.pone.0016877. PMID 21364919
- See also: About EBUS TBNA — http://doi.org/10.1016/j.ejcdt.2013.05.013